CLINICAL TRIAL: NCT01324336
Title: Comparative Pharmacokinetics of a Compounded 6-mercaptopurine Liquid Formulation Preparation and Tablets
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: Midwest Cancer Alliance (Unknown)
Responsible Party: Sponsor
Other Study IDs: 6-MP pharmacokinetic 1
Record Dates: First submitted 2011-03-25; First posted 2011-03-29 (Estimated); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: ALL; acute lymphoblastic leukemia; 6-Mercaptopurine; Pediatric
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Mercaptopurine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 4-17 years, receiving 6-MP
  Interventions: Drug: 6-Mercaptopurine

INTERVENTIONS:
Drug: 6-Mercaptopurine — 75 mg/m2/dose/day
  Other Names: 6-MP

SUMMARY:
The purpose of this study is to compare the pharmacokinetics of a routinely used compounded liquid formulation of 6-mercaptopurine (6-MP) with commercially available tablets in patients who are receiving treatment with 6-MP as part of their clinical treatment for acute lymphoblastic leukemia (ALL).

ELIGIBILITY:
Inclusion Criteria:

* Patients ages 4-17 years of age who are receiving maintenance chemotherapy treatment for ALL with 6-MP will be included.

Exclusion Criteria:

* Inability to have blood drawn for the screening lab tests
* Received methotrexate or folate supplement within the last 24 hours
* Pregnant or lactating females
* Inability to swallow a pill
* Hemoglobin less or equal to 8 gm/dl
* Presence of significant co-morbid illness that makes child ineligible as deemed by the investigator
* Weight < or = 16 kg

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients ages 4-17 years of age who are receiving maintenance chemotherapy treatment for ALL with 6-MP will be included
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2011-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of 6-MP | 8 hours post administration
  To compare the pharmacokinetics of a routinely used compounded liquid formulation of 6-mercaptopurine (6-MP) with commercially available tablets in patients who are receiving treatment with 6-MP as part of their clinical treatment for acute lymphoblastic leukemia (ALL).

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen A Neville, MD, MS, Principal Investigator — The Children's Mercy Hospitals and Clinics
Locations (1):
- The Children's Mercy Hospital, Kansas City, Missouri, United States